CLINICAL TRIAL: NCT05570006
Title: A Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of ABBV-668 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Study of ABBV-668 Oral Capsules to Assess Adverse Events and Change in Disease Activity in Adult Participants With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-446; 2022-501263-41-00 (Other: EU CT)
Record Dates: First submitted 2022-10-05; First posted 2022-10-06 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; ABBV-668
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABBV-668 (Experimental): Participants will receive ABBV-668 twice daily approximately at same time each day for 16 weeks.
  Interventions: Drug: ABBV-668

INTERVENTIONS:
Drug: ABBV-668 — Oral Capsule

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). This study will assess how safe and effective ABBV-668 is in treating adult participants with UC. Adverse events and change in disease activity will be assessed.

ABBV-668 is an investigational drug being developed for the treatment of moderate to severe UC. Approximately 40 adult participants diagnosed with UC will be enrolled in approximately 30 sites globally.

Participants will receive oral capsules of ABBV-668 twice daily for 16 weeks and will undergo a 30 day follow-up period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) for at least 90 days prior to Baseline. Appropriate documentation of biopsy results consistent with the diagnosis of UC in the assessment of the Investigator, must be available.
* Participant meets the following disease activity criteria: Active UC with an Adapted Mayo score of 5 to 9 points and endoscopic subscore of 2 to 3 (confirmed by central review).
* Demonstrated inadequate response to, loss of response to, or intolerance to at least one of the following: oral aminosalicylates, corticosteroids, immunosuppressants and/or targeted immunomodulators (including biologics and non-biologics)

Exclusion Criteria:

* Current diagnosis of crohn's disease (CD) or inflammatory bowel disease-unclassified (IBD-U).
* Extent of inflammatory disease limited to the rectum as assessed by screening endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- United States (18):
  - Gastro SB /ID# 249271, Chula Vista, California
  - Ctr for Advanced Gastroenterol /ID# 249226, Maitland, Florida
  - Atlantic Medical Research /ID# 249213, Margate, Florida
  - Endoscopic Research, Inc. /ID# 249202, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 249278, Macon, Georgia
  - NYU Langone Long Island Clinical Research Associates /ID# 250075, Lake Success, New York
  - Columbia University Medical Center /ID# 250189, New York, New York
  - Lenox Hill Hospital /ID# 250008, New York, New York
  - Atrium Health /ID# 249273, Charlotte, North Carolina
  - Options Health Research, LLC /ID# 249216, Tulsa, Oklahoma
  - University of Pennsylvania /ID# 250012, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute d/b/a AHN Research Institute /ID# 250079, Pittsburgh, Pennsylvania
  - University of Pittsburgh MC /ID# 250071, Pittsburgh, Pennsylvania
  - Gastroenterology Associates, P.A. of Greenville /ID# 249217, Greenville, South Carolina
  - Quality Medical Research /ID# 251125, Nashville, Tennessee
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 249208, Garland, Texas
  - Baylor College of Medicine /ID# 249203, Houston, Texas
  - Southern Star Research Institute, LLC /ID# 249212, San Antonio, Texas
- Belgium (4):
  - UZ Gent /ID# 248605, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 248607, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 248598, Leuven, Vlaams-Brabant
  - Groupe Sante CHC - Clinique du MontLegia /ID# 248928, Liège
- France (4):
  - CHU Montpellier - Hopital Saint Eloi /ID# 251876, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 252108, La Tronche, Isere
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord /ID# 251875, St-Priest-en-Jarez, Pays de la Loire Region
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 252357, Neuilly-sur-Seine, Île-de-France Region
- Poland (4):
  - Gastromed Sp. z o.o /ID# 255664, Torun, Kuyavian-Pomeranian Voivodeship
  - Medical Network Sp.z.o.o. WIP Warsaw IBD Point Profesor Kierkus /ID# 255663, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 255667, Sopot, Pomeranian Voivodeship
  - H-T Centrum Medyczne Endoterapia /ID# 255666, Tychy, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-446

RESULTS

PARTICIPANT FLOW:
Groups:
- ABBV-668: Participants received ABBV-668 twice daily for 16 weeks.
Period: Overall Study
Arm/Group | ABBV-668
Started | 30
Received at Least 1 Dose of Study Drug | 30
Completed | 18
Not Completed | 12
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5
Not completed — Other than Specified | 5

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all participants who received at least 1 dose of study drug.
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Endoscopic Improvement
Description: Endoscopic improvement was defined as Mayo endoscopic subscore of 0 or 1. The endoscopic subscore is scored from 0 (Normal appearance mucosa) to 3 (severe disease, spontaneous bleeding, ulceration) with lower scores associated with better health outcomes.
Time Frame: Week 8
Population: The ITT Population consisted of all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
percentage of participants | 16.7 [3.3 to 30.0]
Statistical Analysis 1: Comparison: ABBV-668; Compared to historical placebo; Test type: Superiority; Bayesian method; Difference in proportion = 7.4

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: From the time of first study drug administration until 30 days after the last dose of study drug (Up to approximately 20 weeks)
Population: The Safety Population consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
Participants | 23

3. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  * Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  * Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  * Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical remission per Adapted Mayo Score was defined as SFS ≤ 1 and not higher than Baseline, RBS of 0, and endoscopic subscore ≤ 1. Data are reported for the percentage of participants achieving clinical remission per adapted Mayo score.
Time Frame: Baseline, Week 8
Population: The ITT Population consisted of all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
percentage of participants | 6.7 [0.0 to 15.6]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Response Per Adapted Mayo Score
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical response per Adapted Mayo Score was defined as a decrease from baseline in the overall score of ≥ 2 points and ≥ 30%, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1. Data are reported for the percentage of participants achieving clinical response per adapted Mayo score.
Time Frame: Baseline, Week 8
Population: The ITT Population consisted of all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
percentage of participants | 33.3 [16.5 to 50.2]

5. Secondary Outcome: Percentage of Participants Achieving Clinical Response Per Partial Adapted Mayo Score
Description: The Partial Adapted Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  The overall Partial Adapted Mayo score ranges from 0 to 6 where higher scores represent more severe disease.
  Clinical response per Partial Adapted Mayo Score was defined as a decrease from baseline in the overall score of ≥ 1 points and ≥ 30%, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1. Data are reported for the percentage of participants achieving clinical response per partial adapted Mayo score.
Time Frame: Baseline, Week 8
Population: The ITT Population consisted of all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
percentage of participants | 40.0 [22.5 to 57.5]

6. Secondary Outcome: Percentage of Participants Achieving Endoscopic Remission
Description: Endoscopic remission was defined as Mayo endoscopic subscore of 0. The endoscopic subscore is scored from 0 (Normal appearance mucosa) to 3 (severe disease, spontaneous bleeding, ulceration) with lower scores associated with better health outcomes.
Time Frame: Week 8
Population: The ITT Population consisted of all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-668
Number analyzed (Participants) | 30
percentage of participants | 6.7 [0.0 to 15.6]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection to the end of the study. The median time on follow-up was 144.0 Days.
Description: All-cause mortality and adverse events: all participants who received at least 1 dose of study drug.
Arm/Group | ABBV-668
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-668 (N=30)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ANOGENITAL DYSPLASIA (Gastrointestinal disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 2 (2)
ILEUS (Gastrointestinal disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-668 (N=30)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 6 (6)
NAUSEA (Gastrointestinal disorders) | 4 (4)
ASTHENIA (General disorders) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05570006/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT05570006/SAP_001.pdf